CLINICAL TRIAL: NCT03242902
Title: Improving Sleep Quality, Psychosocial Functioning, and Cancer Related Fatigue With Light Therapy
Brief Title: To Decrease Fatigue With Light Therapy
Acronym: SPARKLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL61017.031.17
Record Dates: First submitted 2017-07-24; First posted 2017-08-08 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: light therapy; cancer related fatigue; sleep quality; biological rhythms
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light intensity 1 (Experimental): The light intervention includes exposure to white light (10.000 lux) at a distance of 45 cm for 30 minutes within the first half hour after awakening during 3 weeks and 4 days. This can be done while engaged in other activities, for example reading the newspaper or eating breakfast.
  Interventions: Device: Light therapy intensity 1
- Light intensity 2 (Experimental): The light intervention includes exposure to white light (10-20 lux) at a distance of 45 cm for 30 minutes within the first half hour after awakening during 3 weeks and 4 days. This can be done while engaged in other activities, for example reading the newspaper or eating breakfast.
  Interventions: Device: Light therapy intensity 2

INTERVENTIONS:
Device: Light therapy intensity 1 — Exposure to white light (10.000 lux) in the morning
  Arms: Light intensity 1
Device: Light therapy intensity 2 — Exposure to white light (10-20 lux) in the morning
  Arms: Light intensity 2

SUMMARY:
Cancer related fatigue (CRF) is one of the most prevalent and distressing long-term complaints reported by (non-) Hodgkin survivors. The SPARKLE study will test the efficacy of two intensities of light therapy on cancer related fatigue. Additionally, it explores possible working mechanisms of light therapy on CRF including improvements in sleep quality, psychosocial variables (depression, anxiety, cognitive complaints, and quality of life), and changes in biological circadian rhythms.

DETAILED DESCRIPTION:
Rationale: Cancer related fatigue (CRF) is one of the most prevalent and distressing long-term complaints reported by (non-)Hodgkin survivors. So far, there is no standard treatment. Some non-pharmacological interventions have shown large effects but show limitations as well, e.g. they are labor intensive. A novel and promising treatment for CRF is exposure to bright white light (BWL) therapy. This low-cost intervention is easy to deliver and has a low burden for professionals as well as for patients.

Objective: To examine the efficacy of BWL therapy as an intervention for CRF. As a secondary aim, this study will explore possible working mechanisms including changes in sleep quality, psychological variables, biological circadian rhythms, sleep-wake cycles, inflammation markers and genotype.

Study design: A multicenter randomized controlled trial will invite participants and allocate them to either a light intensity 1 condition (n=80) or a light intensity 2 condition (n=80). The longitudinal design will include four measurement points: baseline, mid-intervention, post-intervention, and at 3 and 9 months follow-up.

Study population: Hodgkin and diffuse large B-cell lymphoma (DLBCL) survivors fulfilling the clinical criteria of CRF and a survivorship of ≥ 3 years will be invited. Fatigue should not be attributable to a clear somatic cause or treatment for secondary cancer in the past year. Moreover, 25 Hodgkin survivors without CRF will be recruited to explore the association between circadian rhythms and CRF.

Intervention: The light intervention includes exposure to light for 30 minutes within the first half hour after awakening during 3,5 weeks.

Main study parameters/endpoints: The main study parameter in this study is the change in CRF from baseline to post-intervention and at 3 and 9 months follow-up. This will be assessed with the Multidimensional Fatigue Inventory.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation in this study includes completion of a light intervention for 3,5 weeks (30 min each day) and 2 visits (1h) to the treating hospital pre- and post-intervention. The visits aim to provide instructions and equipment and to collect two blood samples. Additionally, 5 saliva samples will be collected by the participant at home pre- and post-intervention. Moreover, participants complete questionnaires (30 min, 4 times) and wear an accelerometer (10d, 4 times and during light therapy) to objectively measure sleep quality and activity. Risks of the light intervention are limited, although there are few known reports of agitation, headache and nausea during the first days of light exposure. Benefits are the use of an easy to administer treatment for one of the most distressing symptoms that participants report.

ELIGIBILITY:
Inclusion Criteria:

* A history of Hodgkin or DLBCL with a survivorship of ≥ 3 years.
* The presence of moderate to severe fatigue symptoms since diagnosis of or treatment for Hodgkin lymphoma or DLBCL.

Exclusion Criteria:

* Fatigue is explained by a somatic factor as defined in the guidelines of chronic fatigue syndrome of the Dutch internists association (NIV). When a somatic cause for fatigue is resolved by stable medication use ≥ 6 months, patients can be included in the current trial.
* Pregnancy (until 3 months postnatal) or women who provide breast feeding
* Extensive surgical operations in the past 3 months.
* Current diagnosis of a psychiatric disorder (e.g. personality disorders, psychosis, bipolar disorder) which would limit participation.
* Diagnosis of and treatment for a secondary malignancy in the past 12 months.
* Presence of photophobia (abnormal intolerance to visual perception of light) or another eye disease that shows symptoms of photophobia (e.g. aniridia, retinitis pigmentosa, glaucoma).
* Current or previous use of light therapy for more than 1 week.
* Current employment in shift work.
* Insufficient knowledge of the Dutch language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Cancer related fatigue | Change from baseline fatigue at end of 3,5 weeks light therapy
  Fatigue is assessed with the Multidimensional Fatigue Inventory
Cancer related fatigue | Change from baseline fatigue at 3 months after light therapy
  Fatigue is assessed with the Multidimensional Fatigue
Cancer related fatigue | Change from baseline fatigue at 9 months after light therapy
  Fatigue is assessed with the Multidimensional Fatigue

SECONDARY OUTCOMES:
Subjective sleep quality | Change from baseline subjective sleep quality at end of 3,5 weeks light therapy
  Subjective sleep quality is assessed with the Pittsburg Sleep Quality Index
Subjective sleep quality | Change from baseline subjective sleep quality at 3 months after light therapy
  Subjective sleep quality is assessed with the Pittsburg Sleep Quality Index
Subjective sleep quality | Change from baseline subjective sleep quality at 9 months after light therapy
  Subjective sleep quality is assessed with the Pittsburg Sleep Quality Index
Objective sleep quality | Change from baseline objective sleep quality at end of 3,5 weeks light therapy
  Objective sleep quality data is assessed by wearing an accelerometer for 10 days
Objective sleep quality | Change from baseline objective sleep quality at 3 months after light therapy
  Objective sleep quality data is assessed by wearing an accelerometer for 10 days
Objective sleep quality | Change from baseline objective sleep quality at 9 months after light therapy
  Objective sleep quality data is assessed by wearing an accelerometer for 10 days
Depression | Change from baseline depression at end of 3,5 weeks light therapy
  Depression is assessed with the Center for Epidemiological Studies - depression scale
Depression | Change from baseline depression at 3 months after light therapy
  Depression is assessed with the Center for Epidemiological Studies - depression scale
Depression | Change from baseline depression at 9 months after light therapy
  Depression is assessed with the Center for Epidemiological Studies - depression scale
Anxiety | Change from baseline anxiety at end of 3,5 weeks light therapy
  Anxiety is assessed with the State Trait Anxiety Inventory-6 items
Anxiety | Change from baseline anxiety at 3 months after light therapy
  Anxiety is assessed with the State Trait Anxiety Inventory-6 items
Anxiety | Change from baseline anxiety at 9 months after light therapy
  Anxiety is assessed with the State Trait Anxiety Inventory-6 items
Quality of life | Change from baseline quality of life at end of 3,5 weeks light therapy
  Quality of life is assessed with the Medical Outcome studies short form (SF-36)
Quality of life | Change from baseline quality of life at 3 months after light therapy
  Quality of life is assessed with the Medical Outcome studies short form (SF-36)
Quality of life | Change from baseline quality of life at 9 months after light therapy
  Quality of life is assessed with the Medical Outcome studies short form (SF-36)
Subjective cognitive complaints | Change from baseline subjective cognitive complaints at end of 3,5 weeks light therapy
  Subjective cognitive complaints assessed with the Medical Outcomes Studies Cognitive functioning.
Subjective cognitive complaints | Change from baseline subjective cognitive complaints at end of 3,5 weeks light therapy
  Subjective cognitive complaints assessed with the MD Anderson Symptom Inventory
Subjective cognitive complaints | Change from baseline subjective cognitive complaints at 3 months after light therapy
  Subjective cognitive complaints assessed with the Medical Outcomes Studies Cognitive functioning
Subjective cognitive complaints | Change from baseline subjective cognitive complaints at 3 months after light therapy
  Subjective cognitive complaints assessed with the MD Anderson Symptom Inventory
Subjective cognitive complaints | Change from baseline subjective cognitive complaints at 9 months after light therapy
  Subjective cognitive complaints assessed with the Medical Outcomes Studies Cognitive functioning
Subjective cognitive complaints | Change from baseline subjective cognitive complaints at 9 months after light therapy
  Subjective cognitive complaints assessed with the MD Anderson Symptom Inventory
Objective cognitive complaints - alertness and sustained attention | Change from baseline objective cognitive complaints at end of 3,5 weeks light therapy
  Objective cognitive complaints are assessed with the Psychomotor Vigilance Task.
Objective cognitive complaints - long-term memory | Change from baseline objective cognitive complaints at end of 3,5 weeks light therapy
  Objective cognitive complaints are assessed with the 15 words test.
Objective cognitive complaints - short-term memory | Change from baseline objective cognitive complaints at end of 3,5 weeks light therapy
  Objective cognitive complaints are assessed with the digit span task.
Cancer worries | Change from baseline cancer worries at end of 3,5 weeks light therapy
  Cancer worries is assessed with the Cancer Worry scale
Cancer worries | Change from baseline cancer worries at 3 months after light therapy
  Cancer worries is assessed with the Cancer Worry scale
Cancer worries | Change from baseline cancer worries at 9 months after light therapy
  Cancer worries is assessed with the Cancer Worry scale
Fatigue catastrophizing | Baseline
  Fatigue catastrophizing is assessed with the Fatigue catastrophizing scale
Self-efficacy | Baseline
  Self-efficacy is assessed with the Self-efficacy Scale 28
Circadian rhythms of cortisol and melatonin | Change from baseline circadian rhythms at end of 3,5 weeks light therapy
  Circadian rhythms of cortisol and melatonin will be determined from saliva samples
Biomarkers of inflammation and genotype | Change from baseline levels of biomarkers at end of 3,5 weeks light therapy
  Biomarkers of inflammation (hsIL-6, sTNF-RII, IL-1RA, hsCRP, vitamin D) and genotype will be determined from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Bleiker, PhD, Principal Investigator — The Netherlands Cancer Institute; Flora van Leeuwen, Prof.dr.ir., Principal Investigator — The Netherlands Cancer Institute; Laurien Daniels, PhD, MD, Principal Investigator — Leiden University Medical Center
Locations (9):
- Netherlands (9):
  - Radboudumc, Nijmegen, Gelderland
  - Netherlands Cancer Institute, Amsterdam, North Holland
  - VUmc, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Admiraal de Ruyter ziekenhuis, Goes
  - Haga ziekenhuis, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Starreveld DEJ, Daniels LA, Valdimarsdottir HB, Redd WH, de Geus JL, Ancoli-Israel S, Lutgendorf S, Korse CM, Kieffer JM, van Leeuwen FE, Bleiker EMA. Light therapy as a treatment of cancer-related fatigue in (non-)Hodgkin lymphoma survivors (SPARKLE trial): study protocol of a multicenter randomized controlled trial. BMC Cancer. 2018 Sep 10;18(1):880. doi: 10.1186/s12885-018-4746-2. PMID 30200906